CLINICAL TRIAL: NCT06269783
Title: Dual-process Mechanisms of Action for sipIT Intervention Effects in Patients With Urolithiasis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, David Conroy, Bickner Chair of Kinesiology and Professor of Kinesiology, School of Kinesiology, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00022968; R01DK124469 (NIH)
Record Dates: First submitted 2024-02-13; First posted 2024-02-21 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Kidney Stone; Urolithiasis; Nephrolithiasis
MeSH Terms: conditions — Kidney Calculi; Urolithiasis; Nephrolithiasis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- sipIT (Experimental): Participants will receive an educational handout about physical activity, a connected water bottle with its companion mobile application. For months 1-3, participants will receive lapse-contingent reminders to drink delivered by text message.
  Interventions: Behavioral: sipIT

INTERVENTIONS:
Behavioral: sipIT — Automated and manual fluid tracking system with just-in-time reminder messages to support fluid intake habit formation.

SUMMARY:
The purpose of this study is to clarify the fundamental processes underlying behavior change, maintenance, and adherence during and after a 3-month fluid intake intervention period.

DETAILED DESCRIPTION:
The study is a six-month ecological momentary assessment study of patients using the mini-sipIT intervention for 3 months, with weekly assessments of motivation and life events or stressors that disrupt routines during the 3-month intervention period, and monthly assessments of motivation and life events or stressors that disrupt routines in the three months following the end of intervention (months 4-6). The mini-sipIT intervention includes automated and manual tracking of fluid intake and lapse-contingent reminders to drink.

ELIGIBILITY:
Inclusion Criteria:

* Previous diagnosis of symptomatic kidney stone in the past 5 years,
* Age 18 or older,
* Own an iOS or Android smart phone,
* Proficient in English,
* Capable of providing informed consent,
* Willing to use the water bottle and companion app & receive text message reminders for 3 months,
* Live in continental US.

Exclusion Criteria:

* Pregnant or planning to become pregnant during the next 6 months,
* Concurrently participating in other study involving fluid intake or diet,
* Plan to have surgery in the next 6 months,
* Co-morbidities that preclude high fluid intake (congestive heart failure, end-stage renal disease, chronic hyponatremia), or
* Active medical treatments that would impair protocol compliance.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 153 (Actual)
Dates: Start 2024-01-10 (Actual); Primary Completion 2025-02-12 (Actual); Study Completion 2025-05-29 (Actual)

PRIMARY OUTCOMES:
Urine volume (intervention) | from baseline to the end of the intervention period (3 months)
  Change in urine volume

SECONDARY OUTCOMES:
Urine volume (maintenance) | from the end of the intervention period (3 months) to the maintenance change at 6 months
  Change in urine volume

CONTACTS AND LOCATIONS:
Locations (1):
- The Pennsylvania State University, University Park, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No